CLINICAL TRIAL: NCT03788954
Title: Effect of Kinesiotaping on Wrist Kinematics and Functional Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Gürhan KARAKAYA (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Mehmet Gürhan KARAKAYA, Principal investigator, Head of Neurological Rehabilitation Department, Pt. PhD. Prof., Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18/066
Record Dates: First submitted 2018-12-25; First posted 2018-12-28 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Wrist Injuries; Kinematics; Functional Performance
Keywords: Range of motion; Hand injuries; Biomechanics; Rehabilitation
MeSH Terms: conditions — Wrist Injuries; Hand Injuries

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kinesiotaping on FCU (Active Comparator): Muscle fasilitation and Fascia Correction techniques of Kinesiotaping on m. flexor carpi ulnaris.
  Interventions: Other: Kinesiotaping
- Kinesiotaping on ECR (Active Comparator): Muscle fasilitation and Fascia Correction techniques of Kinesiotaping on m. extensor carpi radialis.
  Interventions: Other: Kinesiotaping
- Plasebo Kinesiotaping on FCU (Placebo Comparator): Same kinesiotape used on m. flexor carpi ulnaris without any taping techniques.
  Interventions: Other: Kinesiotaping
- Plasebo Kinesiotaping on ECR (Placebo Comparator): Same kinesiotape used on m. extensor carpi radialis without any taping techniques.
  Interventions: Other: Kinesiotaping

INTERVENTIONS:
Other: Kinesiotaping — Kinesio tape (KT) is the original elastic adhesive tape for injury prevention, rehabilitation, and performance enhancement. Kinesio Tape is latex-free, hypoallergenic and wearable for days at a time. It has been shown to be clinically effective in joint range of motion promotion,increasing muscle activity and functional performance.

SUMMARY:
This study perform to investigate the immediate effects of kinesiotaping and plasebo kinesiotaping on Dart Throwing Motion (DTM) angle and functional performance scores of wrist in healthy subjects.

DETAILED DESCRIPTION:
Kinesiotape which created by Kenzo Kase in 1976, is a thin and elastic taping material similar to the structural properties and flexibility of human skin without limiting joint movements. In this study, kinesiotape will apply to the wrist extensor and flexor muscles using the functional correction and muscle facilitation techniques. Also placebo taping will apply on the same muscles with same kinesiotape without any stretching or positioning. A total of 4 applications including kinesiotaping and placebo taping will perform randomly in 4 consecutive days.

For each subject; A total of 5 separate evaluations will perform on the first day (without taping) and following 4 consecutive days (flexor carpi ulnaris muscle kinesiotaping, extensor carpi radialis muscle kinesiotaping, flexor carpi ulnaris muscle placebo kinesiotaping, extensor carpi radialis muscle placebo kinesiotaping). Between the taping and evaluation of the subjects will wait for 30 minutes.

There are several studies evaluating wrist movements performed in one plane with different methods. The Dart Throwing Motion (DTM) is the most commonly used wrist pattern in daily life and includes the entire oblique movement from radial extension to ulnar flexion.

The aim of this study is to investigate the effects of kinesio taping on the kinematics and functional performance of healthy wrist. This study will be prospective, double-blind, randomized, placebo-controlled and crossover.

We did not find any study including fascia correction kinesiotaping for DTM pattern.

The therapists who works in this area will have an advantage in the rehabilitation programs to know the effects of the muscle facilitation and fascia correction techniques kinesiotaping on wrist kinematics via DTM and wrist functional performance.

Also, we believe that our study will guide different professional groups working on technological rehabilitation with measurement techniques and evaluation methods.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form and participated in all stages of the study
* Being in the age range of 18-25
* Being right-handed

Exclusion Criteria:

* Having physical, mental disability (vision, hearing, etc.) which may affect participation in the study
* Presence of a history of congenital or acquired orthopedic, neurological, or rheumatic disease that may impair joint range and / or function of the hand and wrist
* Having a history of trauma requiring medical, conservative and surgical treatment for the application area in the last 6 months
* Presence of skin lesions (burns, cellulite, vesicles, bulla, pisoriasis, open / closed wound, scar, active infection, malignancy, etc.) in the application area.
* Excessive skin reaction to applications
* The problem of hirsutism to the extent of preventing the kinesiotaping in the application area.
* Dart sports experience as amateur or professional
* To have consumed alcohol, pharmaceutical substance until 24 hours before the evaluation
* Using anabolic substance
* To have theoretical and practical experience in Kinesio taping
* Being obese

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-27 (Actual)

PRIMARY OUTCOMES:
Change of wrist range of motion. | Change of wrist DTM from baseline at the end of 30 minutes of each kinesiotaping intervention.
  Change of wrist dart throwing motion (DTM- radial extansion to ulnar flexion movement of wrist) angle.

SECONDARY OUTCOMES:
Change of wrist functional performance. | Change of MMDT scores from baseline at the end of 30 minutes of each kinesiotaping intervention.
  Change of functional performance of wrist (The Minnesota Manual Dexterity Test - MMDT).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Muğla Sıtkı Koçman University, Muğla, Menteşe
  - Mugla Sıtkı Koçman University, Muğla

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oruk DO, Karakaya MG, Yenisehir S, Karakaya IC. Effect of Kinesio taping on wrist kinematics and functional performance: A randomized controlled trial. J Hand Ther. 2023 Jan-Mar;36(1):3-12. doi: 10.1016/j.jht.2021.09.005. Epub 2021 Oct 27. PMID 34756489